CLINICAL TRIAL: NCT03937557
Title: The Analysis of Hair Count in Healthy Taiwanese Persons by Trichoscope
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chu Gong Yau, Dermatologist, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20190202R
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Dermatosis
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- men's hair count (Active Comparator)
  Interventions: Diagnostic Test: photofinder levicam
- women's hair count (Placebo Comparator)
  Interventions: Diagnostic Test: photofinder levicam

INTERVENTIONS:
Diagnostic Test: photofinder levicam — Exam frontal, bilateral Temporal and occipital scalp by photofinder levicam and compare the pros and cons with the data from scalp biopsy.

SUMMARY:
Horizontal sectioning of scalp biopsy is a better method for evaluating hair disorders than vertical sectioning because it enables the quantitative examination of hair follicles at different stages. Without having the quantitative data of normal scalp hair counts as controls, it is impossible to evaluate scalp biopsies for hair disorders. In recent years, trichoscope is more popular in analysis of hair disease. It is less invasive and simple. The aim of this study is to understand the pros and cons of trichoscpoe.

ELIGIBILITY:
Inclusion Criteria:

* 20-50y/o adults without any scalp disorder

Exclusion Criteria:

* adults with any scalp disorder

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-05 (Estimated); Primary Completion 2020-04-05 (Estimated); Study Completion 2020-04-22 (Estimated)

PRIMARY OUTCOMES:
Average number of hairs | 1 year
  Exam frontal, bilateral Temporal and occipital scalp by photofinder levicam

SECONDARY OUTCOMES:
Average hair shaft thickness | 1 year
  Exam frontal, bilateral Temporal and occipital scalp by photofinder levicam
Amount of Single, double and riple follicular unit | 1year
  Exam frontal, bilateral Temporal and occipital scalp by photofinder levicam
Amount of Empty hair follicles | 1 year
  Exam frontal, bilateral Temporal and occipital scalp by photofinder levicam

IPD SHARING:
Plan to Share IPD: No